CLINICAL TRIAL: NCT03457506
Title: Intra-individual Patient-based Comparison of Conventional and Digital PET/CT Scanners
Brief Title: Intra-individual Comparison of Conventional and Digital PET/CT Scanners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isala (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Piet Jager, Principal Investigator, Isala
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL52329.075.15
Record Dates: First submitted 2017-12-05; First posted 2018-03-07 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer; Lung Cancer; Esophageal Cancer; Miscellaneous Neoplasm
Keywords: Cancer; Digital pet; Conventional pet
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Esophageal Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: All included patients will have two PET scans, one on the conventional PET (Ingenuity TF, Philips Healthcare) and one on the digital PET (Vereos, Philips Healthcare). The order of the two PET scans will differ per patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergo a digital PET/CT (Other): Single arm prospective study of paired PET scans. Patients who are referred to the nuclear medicine department to undergo a PET scan, will undergo a PET/CT scan on the conventional scanner as well as the digital PET/CT scanner.
  Interventions: Diagnostic Test: Digital PET/CT scan

INTERVENTIONS:
Diagnostic Test: Digital PET/CT scan — The digital PET/CT scan will be acquired before or after the conventional PET/CT scan.

SUMMARY:
In this study, the investigators will analyze the impact of digital PET/CT on the final diagnostic conclusion of the scan in patients with lung cancer, breast cancer, esophageal cancer and a group of mescellaneous cancers.

DETAILED DESCRIPTION:
There will be a single injection of the PET radiopharmaceutical FDG, followed by a conventional PET/CT scan and a digital PET scan, in this order or vice versa.

ELIGIBILITY:
Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* referred to Isala for a clinically indicated FDG-PET/CT scan
* suspected or proven lung cancer, esophageal cancer, breast cancer or miscellaneous cancer, either as a primary diagnosis or follow-up study
* signed informed consent

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* age < 18 years
* incapacitated adults
* prisoners
* pregnant patients
* unable to undergo two consecutive PET/CT scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Diagnostic outcome of the PET/CT study | approximately 2 hours

SECONDARY OUTCOMES:
PET image quality | approximately 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pieter L Jager, MD PhD, Principal Investigator — p.l.jager@isala.nl
Locations (1):
- Isala, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koopman D, Jager PL, Slump CH, Knollema S, van Dalen JA. SUV variability in EARL-accredited conventional and digital PET. EJNMMI Res. 2019 Dec 10;9(1):106. doi: 10.1186/s13550-019-0569-7. PMID 31823097

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/06/NCT03457506/Prot_SAP_000.pdf